CLINICAL TRIAL: NCT06439992
Title: Beta Amyloid PET Imaging for Alzheimer Disease: [18F]-Fluselenamyl (Alternative Vehicle) Comparison With [11C]-PIB (FSA-PIB AD)
Brief Title: Beta Amyloid PET Imaging for Alzheimer Disease With [18F]-Fluselenamyl
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology and Neurological Surgery, Washington University School of Medicine
Other Study IDs: FSA-PIB AD
Record Dates: First submitted 2024-04-22; First posted 2024-06-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for future use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Healthy participants with normal cognition will be recruited and receive the following interventions:
  Drug: [18F]-Fluselenamyl. A dosage range of 10 mCi +/- 20% of Fluselenamyl will be injected by a PET-certified medical professional followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]-Pittsburgh Compound ([11C]PIB) A dosage range between 6.0-20.0 mCi is planned. A PET-certified professional will prepare and administer the [11C]-PIB tracer. Participants will receive the PIB injection followed by a 10 ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: 18F-Fluselenamyl
- Participants with mild cognitive impairment: Participants with mild cognitive impairment will be recruited and receive the following interventions:
  Drug: [18F]-Fluselenamyl. A dosage range of 10 mCi +/- 20% of Fluselenamyl will be injected by a PET-certified medical professional followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]-Pittsburgh Compound ([11C]PIB) A dosage range between 6.0-20.0 mCi is planned. A PET-certified professional will prepare and administer the [11C]-PIB tracer. Participants will receive the PIB injection followed by a 10 ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: 18F-Fluselenamyl

INTERVENTIONS:
Drug: 18F-Fluselenamyl — Participants will receive a single intravenous bolus injection of 10 mCi ± 20% of the investigational radiotracer 18F-Fluselenamyl and will undergo an 18F-Fluselenamyl PET/CT scan of the head and neck.
  Other Names: 18F-FSA

SUMMARY:
The purpose of this research study is to determine the safety of a radiotracer 18F-Fluselenamyl using positron emission tomography (PET) imaging.

DETAILED DESCRIPTION:
The investigators will first complete whole-body PET dosimetry studies in healthy adult normal volunteers to calculate the actual radiation dose of each human organ and determine the allowable dose for a human subject when receiving a single dose for a PET scan.

Second, imaging of the brain and neck will be completed in a wide range of ages of healthy adult normal control participants and participants with mild cognitive impairment, both male and females to characterize 18F-Fluselenamyl uptake in the brain, its binding to beta-amyloid plaques, and radiolabeled metabolite will be completed. Amyloid is a protein related to dementia of Alzheimer's disease. 11C-PIB PET imaging and MRI of the brain will also be completed in the same participants and the data will be compared with 18F-Fluselenmayl. 11C-PIB and 18F-Fluselenamyl both bind to beta-amyloid plaques.

Finally, a comparison of the normal control participants to patients with Alzheimer's disease will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, any race
* Age ≥ 18 years
* Healthy volunteers or volunteers with Alzheimer's disease

Exclusion Criteria:

* Has hypersensitivity to 18F-Fluselenamyl or any of its excipients ;
* Has hypersensitivity to 11C-PIB or any of its excipients ;
* Incapable of providing written informed consent or lacking a legally authorized representative (LAR) to provide informed consent ;
* Unwilling or unable to undergo PET scans tracer injections ;
* Unwilling or unable to undergo MRI (Aim 2 and Aim 3)
* Any condition that, in the Investigator's opinion, could increase the risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data (e.g., renal or liver failure, advanced cancer);
* Women who are currently pregnant or breast-feeding;
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: Dosimetry group - 8 healthy adult normal volunteers (4 M, and 4 F) will undergo whole-body PET/CT imaging to assess the safety, dosimetry, and metabolism of 18F-FSA.
  Aim 2: Proof of Concept group - 36 participants (18 healthy and 18 participants with mild cognitive impairment) will undergo 18F-FSA imaging of the brain and neck, 11C-PIB imaging of the brain and neck, MRI, and Cognitive testing.
  Aim 3: Performance group- Aim 2 participants will be invited for additional imaging.
  Aim 3A- 10 participants from Aim 2 will undergo repeat 18F-FSA imaging ~ 1 month after baseline imaging
  Aim 3B- 18 participants from Aim 2 will have a longitudinal follow-up visit ~ 18 months after the initial study. They will undergo repeat 18F-FSA, 11C-PIB, MRI, and Cognitive testing.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of the new formulation of Fluselenamy PET Imaging in 8 healthy adult normal volunteers. | Through study completion, an average of 1 year
  Whole-body PET/CT images (skull vertex to proximal thighs) will be obtained in 8 healthy volunteers (4 males and 4 females) for up to a maximum of 4.5 hours immediately following intravenous (IV) injection of 10 mCi ± 20% of [18F]-Fluselenamyl (dosage range calculated from rodent dosimetry data extrapolated to humans).
  The primary outcome measure is to quantify each organ's radiation exposure (rad/mCi).
PET imaging of [18F]-Fluselenamyl in healthy normal control participants and participants with mild cognitive impairment. | Through study completion, an average of 2 years
  To assess the sensitivity of [18F]-Fluselenamyl to image Amyloid beta in the setting of mild cognitive impairment, and conduct a comparative analysis of PET imaging data using [11C]-PIB imaging in the same participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD., PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States